CLINICAL TRIAL: NCT04948723
Title: Insufficient Awareness and Vaccination Practices for Inflammatory Bowel Disease Patients in China: A Multi-center Survey of Chinese Gastroenterologists
Brief Title: Vaccination Practices for Inflammatory Bowel Disease Patients in China With Gastroenterologists
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Ruijin Hospital (Other); Zhujiang Hospital (Other); Army Medical University, China (Other); Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Lishui Municipal Central Hospital, the Fifth Affiliated Hospital of Wenzhou Medical University (Unknown); Shaoxing Shangyu People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-089
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel diseases， vaccination
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the current study was to evaluate the knowledge of Chinese gastroenterologists on vaccinating patients with IBD under the assistance of Chinese Crohn's & Colitis Foundation. The Chinese Crohn's & Colitis Foundation (CCCF) is the first nonprofit,volunteer-driven foundation specifically for patients with IBD in China.It has been joined by IBD specialists at various hospitals in China.

DETAILED DESCRIPTION:
The questionnaire contained questions regarding the respondents'information, including their gender, years in practice, clinical specialty,and source of knowledge on immunization practices. The questionnaire mainly contained three sections: knowledge of vaccinations for hepatitis A virus (HAV), HBV, and varicella; current vaccination practices for the IBD group; and reasons for not recommending these vaccinations to patients with IBD. The questionnaire composed of 13 items specifically on the three vaccinations mentioned above for immunosuppressed patients with IBD. All questions were conducted based on recognized guidelines and were reviewed by 18 IBD experts. The questionnaire captured the frequency with which the respondents assessed patients with IBD for anti-HAV/hepatitis B surface antigen (HBsAg), hepatitis B core antibody, and hepatitis B surface antibody/ anti-HAV levels, and acquired infection and immunization histories. Whether the respondents recommended these three vaccines to the IBD group before treatment was also elicited.

ELIGIBILITY:
Inclusion Criteria:

* gastroenterologists were members of tertiary hospitals

Exclusion Criteria:

* pediatricians were excluded, as were retired gastroenterologists and those currently in training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An email with a quick response code (QRC) was sent to CCCF-affiliated gastroenterologists specializing in IBD between July 2017 and August 2017
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
vaccination practices | between July 2017 and August 2017
  The questionnaire mainly contained three sections: knowledge of vaccinations for hepatitis A virus (HAV), HBV, and varicella; current vaccination practices for the IBD group; and reasons for not recommending these vaccinations to patients with IBD. The questionnaire captured the frequency with which the respondents assessed patients with IBD for anti-HAV/hepatitis B surface antigen (HBsAg), hepatitis B core antibody, and hepatitis B surface antibody/ anti-HAV levels, and acquired infection and immunization histories.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Study Director — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Shuyan Li, Zhejiang, Hangzhou, China